CLINICAL TRIAL: NCT00056160
Title: A Multicenter, Randomized, Parallel-Group, Double-blind, Placebo-controlled Study of CC-5013 Plus Dexamethasone Versus Dexamethasone Alone in Previously Treated Subjects With Multiple Myeloma
Brief Title: CC-5013 Plus Dexamethasone Versus Dexamethasone Alone in Previously Treated Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-MM-009
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Results first posted 2010-03-03 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Refractory and Relapsed; Revlimid; CC5013
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CC-5013/Dex (Experimental): CC-5013 (lenalidomide) plus oral high-dose dexamethasone
  Interventions: Drug: CC-5013; Drug: Dexamethasone
- Placebo/Dex (Experimental): Placebo, identical in appearance to CC-5013 (lenalidomide), plus oral high-dose dexamethasone
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: CC-5013 — Subjects in the CC-5013/Dex treatment group took 25 mg of lenalidomide orally once daily on Days 1 to 21 and a matching placebo capsule once daily on Days 22 to 28 of each 28-day cycle.
  Other Names: lenalidomide; Revlimid
  Arms: CC-5013/Dex
Drug: Dexamethasone — Subjects in the CC-5013/Dex and Placebo/Dex treatment groups took 40 mg of dexamethasone orally once daily on Days 1 to 4, 9 to 12, and 17 to 20 of each 28-day cycle for the first 4 cycles of therapy. Beginning with Cycle 5, the dose of dexamethasone was reduced to 40 mg orally once daily on Days 1 to 4 for the remaining cycles.
  Other Names: Decadron

SUMMARY:
Randomized subjects will receive CC-5013 plus high-dose dexamethasone or placebo appearing identical to CC-5013 plus high-dose dexamethasone in 4-week cycles. Each subject will participate in a treatment phase and a follow-up phase.

DETAILED DESCRIPTION:
This was a phase 3, multicenter, double-blind, placebo-controlled, parallel-group study of the efficacy and safety of CC-5013 plus oral pulse high-dose dexamethasone and oral pulse high-dose dexamethasone therapy alone in subjects with relapsed or refractory multiple myeloma. Eligible subjects were randomized in a 1:1 ratio to 1 of 2 treatment groups: Subjects in the CC-5013/Dex treatment group took 25 mg of CC-5013 orally once daily on Days 1 to 21 and a matching placebo capsule once daily on Days 22 to 28 of each 28-day cycle; Subjects in the Placebo/Dex treatment group took 1 placebo capsule on Days 1 to 28 of each 28-day cycle. Subjects in both treatment groups took 40 mg of dexamethasone orally once daily on Days 1 to 4, 9 to 12, and 17 to 20 of each 28-day cycle for the first 4 cycles of therapy. Beginning with Cycle 5, the dose of dexamethasone was reduced to 40 mg orally once daily on Days 1 to 4 for the remaining cycles.

ELIGIBILITY:
Inclusion Criteria:

* Prior or current diagnosis Durie-Salmon stage II or III multiple myeloma.
* No more than 3 previous anti-myeloma regimens
* No high-dose dexamethasone (total monthly dose of dexamethasone greater than 200 mg) within 6 months of study randomization.
* Measurable levels of myeloma paraprotein in serum or urine (24-hour collection sample).

Exclusion Criteria:

* Prior development of disease progression during high-dose dexamethasone containing therapy.
* Laboratory abnormalities: Absolute neutrophil count less than 1,000 cells/mm cubed
* Laboratory abnormalities: Platelet count less than 75,000/mm cubed
* Laboratory abnormalities: Serum creatinine greater than 2.5 mg/dL
* Laboratory abnormalities: Serum glutamic oxaloacetic transaminase (SGOT, aspartate transaminase [AST]) or serum glutamic pyruvic transaminase (SGPT, alanine transaminase [ALT])greater than 3.0 x upper limit of normal
* Laboratory abnormalities: Serum total bilirubin greater than 2.0 mg/dL
* Prior history of malignancies other than multiple myeloma unless the subject has been free of the disease for greater than or equal to 5 years.
* Known hypersensitivity to thalidomide or dexamethasone.
* Development of a desquamating rash while taking thalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2005-11-01 (Actual); Study Completion 2008-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (49):
- United States (44):
  - Clinical Research Consultants, Inc., Hoover, Alabama
  - City of Hope National Medical Center, Duarte, California
  - UCLA School of Medicine, Los Angeles, California
  - UCSF California, San Francisco, California
  - Stanford University Medical Center, Division of Hematology, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Mayo Clinic- Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Oncology Hematology Consultants, Sarasota, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Northwestern University Med Ctr, Chicago, Illinois
  - Rush Cancer Institute Section of Hematology, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana Cancer Research Institute, Indianapolis, Indiana
  - University of Iowa Hospital Clinic, Iowa City, Iowa
  - Ocshner Clinical Foundation, New Orleans, Louisiana
  - Johns Hopkins Medicine Department of Oncology, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University Of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University School of Medicine- Sherman Cancer Center, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - MBCCOP Our Lady of Mercy Cancer Center New York Medical College, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic Myeloma Program, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Kaiser Permanente Northwest Region Center for Health Research, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Charleston Hematology/Oncology P.A., Charleston, South Carolina
  - Medical University of SC, Charleston, South Carolina
  - South Carolina Oncology Group, West Columbia, South Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital/BMT Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - Dalhousie University, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
  - Hospital Charles LeMoyne, Greenfield Park, Quebec
  - McGill University, Montreal, Quebec

REFERENCES:
- [Result] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763
- [Derived] San-Miguel JF, Dimopoulos MA, Stadtmauer EA, Rajkumar SV, Siegel D, Bravo ML, Olesnyckyj M, Knight RD, Zeldis JB, Harousseau JL, Weber DM. Effects of lenalidomide and dexamethasone treatment duration on survival in patients with relapsed or refractory multiple myeloma treated with lenalidomide and dexamethasone. Clin Lymphoma Myeloma Leuk. 2011 Feb;11(1):38-43. doi: 10.3816/CLML.2010.n.120. PMID 21273172
- [Derived] Zangari M, Tricot G, Polavaram L, Zhan F, Finlayson A, Knight R, Fu T, Weber D, Dimopoulos MA, Niesvizky R, Fink L. Survival effect of venous thromboembolism in patients with multiple myeloma treated with lenalidomide and high-dose dexamethasone. J Clin Oncol. 2010 Jan 1;28(1):132-5. doi: 10.1200/JCO.2009.23.0169. Epub 2009 Nov 9. PMID 19901114
- [Derived] Wang M, Dimopoulos MA, Chen C, Cibeira MT, Attal M, Spencer A, Rajkumar SV, Yu Z, Olesnyckyj M, Zeldis JB, Knight RD, Weber DM. Lenalidomide plus dexamethasone is more effective than dexamethasone alone in patients with relapsed or refractory multiple myeloma regardless of prior thalidomide exposure. Blood. 2008 Dec 1;112(12):4445-51. doi: 10.1182/blood-2008-02-141614. Epub 2008 Sep 17. PMID 18799726
- See also: Link to CSR synopsis — http://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/clinical-study-report-csr-synopses/purposes-of-posting-clinical-study-report-csr-synopses

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects in the Placebo/Dex treatment group did not continue participation beyond the period "Up To Unblinding (07 Jun 2005"). Only subjects in the CC-5013/Dex treatment group participated in the period "Extended Follow-up Cutoff (23 Jul 2008)".
Pre-assignment Details: Only subjects in the CC-5013/Dex treatment group participated in the period "Extended Follow-up Cutoff (23 Jul 2008)". Data for the period "Extended Follow-up Cutoff (23 Jul 2008)" subsumes data for the period "Up To Unblinding (07 Jun 2005)".
Period: Up to Unblinding (07 Jun 2005)
Arm/Group | CC-5013/Dex | Placebo/Dex
Started | 177 | 176
Completed | 64 | 13
Not Completed | 113 | 163
Not completed — Adverse Event | 35 | 18
Not completed — Progression of disease | 57 | 124
Not completed — Lack of Efficacy | 3 | 5
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Death | 2 | 1
Not completed — Other | 8 | 7
Period: Extended Follow-up Cutoff (23 Jul 2008)
Arm/Group | CC-5013/Dex | Placebo/Dex
Started | 177 | 0
Completed | 6 | 0
Not Completed | 171 | 0
Not completed — Adverse Event | 44 | 0
Not completed — Progression of disease | 87 | 0
Not completed — Lack of Efficacy | 3 | 0
Not completed — Withdrawal by Subject | 11 | 0
Not completed — Death | 5 | 0
Not completed — Other | 21 | 0
Period: Final Follow-up
Arm/Group | CC-5013/Dex | Placebo/Dex
Started | 6 | 0
Completed | 0 | 0
Not Completed | 6 | 0
Not completed — Transferred into expanded access study. | 3 | 0
Not completed — Transferred into RevAssist Program | 2 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CC-5013/Dex | Placebo/Dex | Total
Number analyzed (Participants) | 177 | 176 | 353
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 103 | 197
  >=65 years | 83 | 73 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.84) | 62.5 (9.81) | 62.9 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 72 | 143
  Male | 106 | 104 | 210
Region of Enrollment [Number; unit: participants]
  United States | 142 | 150 | 292
  Canada | 35 | 26 | 61

OUTCOME MEASURES:

1. Primary Outcome: Time to Tumor Progression (TTP)
Description: Time to progression (TTP) was calculated as the time from randomization to the first documentation of progressive disease based on the myeloma response determination criteria developed by Bladé et. al., Br J Haematol 1998; 102:1115-1123.
Time Frame: 60 weeks (median Time To Progression of CC-5013/Dex treatment group)
Population: Analysis conducted on the Intent-To-Treat (ITT) Population. The ITT Population was defined as all subjects randomized.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | CC-5013/Dex | Placebo/Dex
Number analyzed (Participants) | 177 | 176
Weeks | 60.1 [41.1 to 80.0] | 20.1 [16.1 to 21.1]

2. Secondary Outcome: Overall Survival
Description: Overall survival was calculated as the time from randomization to death from any cause.
Time Frame: 170 weeks (median overall survival of CC-5013/Dex treatment group)
Population: Analysis conducted on the Intent-To-Treat (ITT) Population. The ITT Population was defined as all subjects randomized.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | CC-5013/Dex | Placebo/Dex
Number analyzed (Participants) | 177 | 176
Weeks | 170.1 [142.1 to 204.9] | 136.4 [104.1 to 176.9]

3. Secondary Outcome: Myeloma Response
Description: The overall confirmed response that was maintained for ≥6 weeks. Complete Response (CR):Disappearance of monoclonal paraprotein. Remission Response (RR):75-99% reduction in monoclonal paraprotein/90-99% reduction in 24-hr urinary light chain excretion. Partial Response (PR):50-74% reduction in monoclonal paraprotein/50-89% reduction in 24-hr urinary light chain excretion. Stable Disease (SD):Criteria for PR or PD not met. Plateau Phase:If PR, stable monoclonal paraprotein (within 25% above or below nadir)/stable soft tissue plasmacytomas. Progressive Disease (PD):Disease worsens.
Time Frame: Up to Unblinding (07 Jun 2005)
Population: Analysis conducted on the Intent-To-Treat (ITT) Population. The ITT Population was defined as all subjects randomized. Results reported (Response) are numbers of subjects.
Measure: Number; unit: Participants
Arm/Group | CC-5013/Dex | Placebo/Dex
Number analyzed (Participants) | 177 | 176
Participants | 107 | 34

4. Secondary Outcome: Time to First Worsening of Eastern Cooperative Oncology Group (ECOG) Performance Status Scale (Best Score=0, Fully Active, Able to Carry on All Pre-disease Performance Without Restriction; Worst Score=5, Dead.)
Description: The time to first worsening on the ECOG Performance Scale was calculated as the time from randomization to the date of the first worsening compared to the last ECOG evaluation obtained prior to randomization.
Time Frame: 30 weeks (mean time to first worsening of ECOG performance status for CC-5013/Dex treatment group)
Population: Analysis conducted on the Intent-To-Treat (ITT) Population. The ITT Population was defined as all subjects randomized.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | CC-5013/Dex | Placebo/Dex
Number analyzed (Participants) | 177 | 176
Weeks | 29.9 (30.02) | 15.0 (16.98)

ADVERSE EVENTS:
Time Frame: Up to 254 weeks (median=48 weeks; mean=77 weeks)
Description: Analyses of safety (Serious Adverse Events and Other Adverse Events) were based upon the Safety Population (all subjects who were administered at least one dose of study medication) and include all data available.
Arm/Group | CC-5013/Dex | Placebo/Dex
Serious Adverse Events (participants affected / at risk) | 111/177 | 90/175
Other Adverse Events (participants affected / at risk) | 177/177 | 175/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CC-5013/Dex (N=177) | Placebo/Dex (N=175)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (4) | 1 (1)
ABSCESS INTESTINAL (Infections and infestations) | 0 (0) | 1 (1)
ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ACQUIRED BRONCHOMALACIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 (3) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 2 (3) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 2 (3) | 3 (3)
ANAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 2 (2) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 1 (1) | 0 (0)
APPENDICEAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ARTERIAL THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
ARTERIOSPASM CORONARY (Cardiac disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 2 (2) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 10 (11) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 2 (2) | 0 (0)
AZOTAEMIA (Renal and urinary disorders) | 0 (0) | 1 (1)
BLINDNESS (Eye disorders) | 1 (1) | 0 (0)
BLINDNESS TRANSIENT (Eye disorders) | 1 (1) | 0 (0)
BLOOD BILIRUBIN ABNORMAL (Investigations) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BRONCHIOLOALVEOLAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 4 (4) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CATARACT UNILATERAL (Eye disorders) | 0 (0) | 1 (1)
CATHETER RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CATHETER SITE PAIN (General disorders) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0)
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
CEREBELLAR INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 5 (5) | 1 (1)
CHEST PAIN (General disorders) | 2 (2) | 0 (0)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
CLOSTRIDIUM COLITIS (Infections and infestations) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS PSEUDOMEMBRANOUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
CONVULSIONS (Nervous system disorders) | 0 (0) | 3 (3)
CORONARY ARTERY DISEASE (Cardiac disorders) | 3 (3) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 18 (18) | 6 (6)
DEHYDRATION (Metabolism and nutrition disorders) | 7 (9) | 5 (5)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0)
DELUSION (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DIABETES WITH HYPEROSMOLARITY (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 0 (0)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIVERTICULITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2) | 0 (0)
DYSPNOEA EXACERBATED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
EMPHYSEMATOUS BULLA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ENCEPHALITIS HERPES (Infections and infestations) | 0 (0) | 1 (1)
ENTEROBACTER BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
FANCONI SYNDROME ACQUIRED (Renal and urinary disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATITIS TOXIC (Hepatobiliary disorders) | 0 (0) | 1 (1)
HERPES VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
HYPERAMMONAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0)
HYPERVISCOSITY SYNDROME (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (24) | 1 (1)
INFECTION (Infections and infestations) | 2 (2) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 2 (2) | 0 (0)
INTERSTITIAL PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTRACRANIAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
INTRACRANIAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 1 (1) | 0 (0)
LARGE INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
LEUKAEMIA PLASMACYTIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
LEUKOENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
LIVER FUNCTION TESTS ABNORMAL (Investigations) | 1 (1) | 0 (0)
LOBAR PNEUMONIA (Infections and infestations) | 4 (6) | 1 (1)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
LUNG NODULE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
MAJOR DEPRESSIVE DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 3 (3)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
MYOPATHY STEROID (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 1 (1)
PLASMACYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMOCYSTIS CARINII PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 1 (1)
PNEUMONIA CYTOMEGALOVIRAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA FUNGAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 30 (39) | 15 (17)
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
PULMONARY OEDEMA (Cardiac disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 7 (8) | 6 (8)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 (3) | 2 (2)
RENAL FAILURE (Renal and urinary disorders) | 3 (3) | 5 (5)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0)
RETINAL VEIN OCCLUSION (Eye disorders) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
SEPSIS (Infections and infestations) | 3 (3) | 2 (2)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
SINUSITIS FUNGAL (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 2 (2) | 0 (0)
SKIN DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 2 (2)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
SUBACUTE ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Nervous system disorders) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0)
SUPERIOR VENA CAVAL OCCLUSION (Vascular disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 3 (4) | 1 (1)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 4 (5) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0)
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CC-5013/Dex (N=177) | Placebo/Dex (N=175)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 11 (12) | 15 (18)
ABDOMINAL PAIN (Gastrointestinal disorders) | 20 (27) | 12 (15)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 11 (13) | 10 (12)
AGEUSIA (Nervous system disorders) | 10 (13) | 7 (7)
ANAEMIA (Blood and lymphatic system disorders) | 72 (139) | 37 (44)
ANOREXIA (Metabolism and nutrition disorders) | 35 (39) | 22 (23)
ANXIETY (Psychiatric disorders) | 32 (38) | 20 (22)
APPETITE DECREASED (Metabolism and nutrition disorders) | 21 (25) | 12 (14)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 41 (63) | 35 (51)
ASTHENIA (General disorders) | 43 (59) | 47 (66)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 57 (71) | 38 (40)
BALANCE IMPAIRED (Nervous system disorders) | 10 (11) | 3 (3)
BLOOD CREATININE INCREASED (Investigations) | 9 (13) | 6 (6)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 20 (31) | 15 (25)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 19 (24) | 3 (7)
CATARACT (Eye disorders) | 9 (10) | 1 (1)
CATARACT UNILATERAL (Eye disorders) | 10 (15) | 2 (3)
CELLULITIS (Infections and infestations) | 10 (11) | 3 (3)
CHEST PAIN (General disorders) | 22 (34) | 15 (24)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 17 (18) | 9 (9)
CONFUSIONAL STATE (Psychiatric disorders) | 22 (25) | 14 (16)
CONSTIPATION (Gastrointestinal disorders) | 74 (99) | 35 (43)
CONTUSION (Skin and subcutaneous tissue disorders) | 20 (23) | 13 (15)
COUGH (Respiratory, thoracic and mediastinal disorders) | 53 (91) | 48 (53)
CUSHINGOID (Endocrine disorders) | 12 (13) | 13 (13)
DEEP VEIN THROMBOSIS (Vascular disorders) | 10 (10) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 21 (26) | 9 (10)
DEPRESSION (Psychiatric disorders) | 29 (31) | 19 (19)
DIARRHOEA (Gastrointestinal disorders) | 85 (174) | 53 (85)
DIZZINESS (Nervous system disorders) | 51 (102) | 43 (54)
DRY MOUTH (Gastrointestinal disorders) | 17 (18) | 8 (10)
DRY SKIN (Skin and subcutaneous tissue disorders) | 19 (24) | 10 (13)
DYSGEUSIA (Nervous system disorders) | 34 (37) | 19 (23)
DYSPEPSIA (Gastrointestinal disorders) | 37 (41) | 28 (37)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 12 (12)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 51 (64) | 39 (47)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 16 (21) | 11 (12)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 10 (12) | 6 (6)
FACE OEDEMA (Skin and subcutaneous tissue disorders) | 13 (15) | 13 (13)
FATIGUE (General disorders) | 114 (191) | 105 (164)
FLATULENCE (Gastrointestinal disorders) | 16 (18) | 9 (10)
FLUID RETENTION (Metabolism and nutrition disorders) | 9 (9) | 2 (3)
FLUSHING (Vascular disorders) | 12 (13) | 12 (12)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 10 (13) | 4 (5)
HEADACHE (Nervous system disorders) | 56 (79) | 54 (66)
HERPES SIMPLEX (Infections and infestations) | 15 (22) | 6 (6)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 11 (26) | 9 (9)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 14 (14)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 37 (62) | 24 (28)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 10 (11) | 2 (2)
HYPERTENSION (Nervous system disorders) | 17 (17) | 11 (15)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 17 (22) | 4 (5)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 34 (91) | 12 (17)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 21 (34) | 8 (8)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 9 (11) | 5 (5)
HYPOTENSION (Vascular disorders) | 20 (21) | 5 (5)
INFLUENZA LIKE ILLNESS (General disorders) | 10 (11) | 3 (5)
INSOMNIA (Psychiatric disorders) | 84 (99) | 70 (84)
IRRITABILITY (Psychiatric disorders) | 20 (21) | 11 (11)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 9 (11) | 2 (2)
LETHARGY (General disorders) | 11 (12) | 4 (4)
LEUKOPENIA (Blood and lymphatic system disorders) | 15 (20) | 3 (3)
LIVER FUNCTION TESTS ABNORMAL (Investigations) | 10 (11) | 3 (3)
LOOSE STOOLS (Gastrointestinal disorders) | 13 (14) | 10 (13)
MOOD ALTERATION (Psychiatric disorders) | 5 (6) | 17 (17)
MOOD SWINGS (Psychiatric disorders) | 9 (9) | 4 (4)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 69 (120) | 41 (61)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 9 (11) | 5 (6)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 27 (37) | 29 (31)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (7)
MYALGIA (Musculoskeletal and connective tissue disorders) | 21 (22) | 22 (26)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 7 (8)
NASOPHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 39 (82) | 11 (13)
NAUSEA (Gastrointestinal disorders) | 58 (90) | 55 (79)
NEUROPATHY (Nervous system disorders) | 21 (25) | 12 (13)
NEUTROPENIA (Blood and lymphatic system disorders) | 87 (348) | 12 (22)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 16 (20) | 13 (16)
NOCTURIA (Renal and urinary disorders) | 6 (6) | 10 (11)
OEDEMA (General disorders) | 15 (22) | 18 (22)
OEDEMA PERIPHERAL (General disorders) | 58 (87) | 42 (54)
ORAL CANDIDIASIS (Infections and infestations) | 14 (18) | 10 (11)
ORAL PAIN (Gastrointestinal disorders) | 10 (12) | 1 (1)
PAIN IN LIMB (Musculoskeletal and connective tissue disorders) | 28 (38) | 13 (23)
PAIN (General disorders) | 20 (23) | 19 (25)
PARAESTHESIA (Nervous system disorders) | 24 (31) | 18 (23)
PERIPHERAL NEUROPATHY (Nervous system disorders) | 27 (33) | 19 (23)
PERIPHERAL SWELLING (Musculoskeletal and connective tissue disorders) | 18 (21) | 4 (5)
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 33 (55) | 18 (22)
PNEUMONIA (Infections and infestations) | 23 (31) | 4 (4)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 7 (7)
PRURITUS (Skin and subcutaneous tissue disorders) | 20 (30) | 10 (11)
PYREXIA (General disorders) | 54 (85) | 35 (48)
RASH (Skin and subcutaneous tissue disorders) | 55 (83) | 28 (30)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 5 (6)
RIGORS (General disorders) | 10 (15) | 14 (16)
SINUSITIS (Infections and infestations) | 26 (41) | 11 (14)
SOMNOLENCE (Nervous system disorders) | 10 (10) | 7 (8)
STOMATITIS (Gastrointestinal disorders) | 15 (23) | 14 (15)
SWEATING INCREASED (Skin and subcutaneous tissue disorders) | 19 (21) | 10 (11)
SYNCOPE (Nervous system disorders) | 9 (16) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 45 (83) | 19 (28)
TOOTHACHE (Gastrointestinal disorders) | 10 (11) | 5 (5)
TREMOR (Nervous system disorders) | 36 (44) | 12 (15)
UPPER RESPIRATORY TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 63 (123) | 39 (59)
URINARY FREQUENCY (Renal and urinary disorders) | 11 (13) | 7 (8)
URINARY TRACT INFECTION (Infections and infestations) | 18 (31) | 7 (13)
VISION BLURRED (Eye disorders) | 50 (79) | 30 (56)
VOMITING (Gastrointestinal disorders) | 26 (32) | 22 (24)
WEIGHT DECREASED (Investigations) | 20 (24) | 8 (8)

LIMITATIONS AND CAVEATS:
Analyses for efficacy had data cutoff dates of 07 Jun 2005 and a data cutoff date of 23 Jul 2008 for overall survival. Only safety data were collected for 6 subjects ongoing beyond the 23 Jul 2008 data cutoff date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present the clinical data generated from the study provided that such Investigator shall furnish sponsor with a copy of the proposed publication or presentation at least 60 days in advance of submission, delete any confidential information, and delay submission for up to 90 days to permit the preparation and filing of appropriate intellectual property applications.